CLINICAL TRIAL: NCT02146092
Title: Incentive Spirometry Added to Physiotherapy to Reduce Postoperative Pulmonary Complications After Lung Surgery: A Prospective Blinded Randomized Trial
Brief Title: Incentive Spirometry Added to Physiotherapy to Reduce Postoperative Pulmonary Complications After Lung Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: McMaster Surgical Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SJHH_Spirometry001
Record Dates: First submitted 2014-05-12; First posted 2014-05-23 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Lung Neoplasms; Benign Lung Disease
Keywords: lung resection; incentive spirometry; physiotherapy; quality improvement; outcomes; post operative complications
MeSH Terms: conditions — Lung Neoplasms | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard physiotherapy (Active Comparator): Standard physiotherapy includes routine physiotherapy care as per current institutional standards. This consists of two daily visits by the physiotherapist. During the visits, the patient will be taught deep breathing and will be instructed to practice it 10 times every hour. They are also shown shoulder movements and lung expansion exercises. They will receive a sheet summarizing the exercises for future reference. The patient is discharged from physiotherapy when they are ambulatory, on room air, and able to clear their respiratory secretions independently, although they will be asked to continue the exercises on their own until 30 days from surgery.
  Interventions: Other: Physiotherapy
- Incentive Spirometry (Experimental): Patients in the Incentive Spirometry arm will receive standard physiotherapy care in addition to training and use of an incentive spirometer. The physiotherapy care includes routine care as per current institutional standards.
  They will also receive an incentive spirometer on the first postoperative day and will be taught how to use it with an accompanying instructional sheet for later reference. Teaching will emphasize slow deep breathing, sustained vacuum pressure, and gradual increase in difficulty. Patients will be instructed to use the spirometer 10 times every hour until 30 days after surgery.
  Interventions: Procedure: Incentive spirometry; Other: Physiotherapy

INTERVENTIONS:
Procedure: Incentive spirometry
  Arms: Incentive Spirometry
Other: Physiotherapy — Standard of care exercise training and supervision

SUMMARY:
After any surgery, there is a chance of complications. After lung surgery to remove tumours, there is a particularly high chance of a person developing an infection or needing help breathing, called post operative pulmonary complications. Currently, the risk of these complications is reduced through the completion of light physical and deep breathing exercises and walking around as soon as possible after surgery. Another possible way of helping these patients is to use a small device called an Incentive Spirometer to encourage and measure deep breathing. This study wants to compare how often postoperative pulmonary complications happen after major lung surgery between a group completing the exercises alone and a group using the Incentive spirometer in addition to the exercises. It is hoped that the combined therapy will reduce the amount of time patient must stay in hospital, have fewer complication events and have fewer patients re-admitted back into the hospital after they go home, so that patients overall have better outcomes.

DETAILED DESCRIPTION:
This study is a prospective blinded randomized control trial (RCT) where two arms will be assembled. Consenting eligible patients will be randomized to either the physiotherapy + incentive spirometry (PT+IS-intervention) arm or physiotherapy only (PT-control arm). Patients will be randomized with an equal (1:1) chance of being allocated to either the PT (control) arm or PT+IS (intervention) arm. Both the treating surgeon and data interpreter will be blinded to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at minimum age 18
* Patient must be undergoing pulmonary resection surgery for malignant or benign disease
* Patients must be able to understand English
* Patients must be able to demonstrate aptitude and willingness to comply with describes study procedures

Exclusion Criteria:

* Patients who are unable to read and communicate in English
* Home oxygen usage prior to operation
* Previous pulmonary resection or any thoracic surgery
* Radiological evidence of atelectasis or pneumonitis on preoperative imaging
* Radiological evidence of pleural effusion prior on preoperative imaging
* Prior exposure to pulmonotoxic drugs such as amiodarone or belomycin
* Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Rate of post operative pulmonary complications within 30 days of surgery | 30 days after surgery
  Postoperative pulmonary complications (PPCs) are defined as:
  * Pneumonia requiring treatment with antibiotics
  * Atelectasis requiring pulmonary toilet by bronchoscopy
  * Respiratory failure requiring treatment via mechanical ventilation (invasive or non-invasive)
  * Requirement for home oxygen after surgery, when this was not the case prior to surgery

SECONDARY OUTCOMES:
Duration of oxygen treatment in hospital | 30 days post-surgery
  Use of oxygen therapy required while in hospital
Length of hospital stay | 30 days after surgery
Re-admission to hospital | 30 days
  Re-admission to hospital due to post operative pulmonary complications
Cost effectiveness of spirometry utilization | 30 days after surgery
  Calculated as an aggregate measure considering length of hospital stay, readmission to hospital and cost of treating complications. A cost value will be assigned to each group and compared for cost-benefit relationships

CONTACTS AND LOCATIONS:
Overall Officials: Wael C Hanna, MDCM MBA FRCSC FCCP, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No